CLINICAL TRIAL: NCT05699551
Title: Supervised Exercise as a Therapeutic Strategy for Interstitial Cystitis/Bladder Pain Syndrome
Acronym: IC/BPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00092907
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: exercise; interstitial cystitis; bladder
MeSH Terms: conditions — Cystitis, Interstitial; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise treatment group (Experimental): This group will serve as both their own controls and study subjects for the experimental intervention. They will take surveys to record bladder symptoms and quality of life before undergoing exercise. They will then take the same surveys after exercise and their scores will be compared.
  Interventions: Behavioral: Exercise regimen

INTERVENTIONS:
Behavioral: Exercise regimen — Exercise will take place Monday, Wednesday, and Friday from 12:00-1:00 pm for 6 weeks. Aerobic exercise will consist of walking, beginning with a 10-minute duration, with gradual progression to 20 minutes. Muscle strength, endurance and range-of-motion exercise will then be performed. Muscle strength and endurance training will begin using no weight and performing one set of 6 repetitions. Progression using added resistance in the form of dumbbell weights (1-6 lbs.) and increased sets and repetitions will be applied as Subjects become increasingly fit. For static range of motion exercise, positions will be held for 10-15 seconds in the beginning and increased over time. Exercise will be kept at a moderate level of intensity. Each session will then end with relaxation training.

SUMMARY:
In this study, the efficacy of exercise to improve interstitial cystitis/bladder pain syndrome symptoms and quality of life will be investigated.

DETAILED DESCRIPTION:
Effective treatment for symptoms associated with interstitial cystitis/bladder pain syndrome is a significant clinical challenge due to the lack of insight into disease etiology/pathophysiology, costly and potentially invasive procedures, and a lack of research into potential therapeutics. The primary objective of this study is to determine if a supervised exercise program by a trained exercise physiologist can relieve pain and improve urinary and bladder symptoms in patients with interstitial cystitis/bladder pain syndrome. This has the potential to open enormous future avenues of research, save both patients and the healthcare system cost, and most importantly improve patients' lives. A second objective of this study is to determine if exercise alters depressive symptoms, often a comorbid diagnosis, in patients with interstitial cystitis/bladder pain syndrome. A third objective of this study is to examine urinary markers of inflammation before and after exercise in patients with interstitial cystitis/bladder pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult females (>18 years and <80 years) with a previously established clinical diagnosis of Interstitial cystitis/bladder pain syndrome (IC/BPS) will be eligible to participate
* Must speak English
* The clinical diagnosis of IC/BPS will be based on the recently published American Urological Association Guidelines definition: "An unpleasant sensation (pain, pressure, or discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms for more than six weeks duration, in the absence of infection or other identifiable causes"
* The diagnosis will be confirmed by a urologist who specializes in the treatment of patients with IC/BPS

Exclusion Criteria:

* Study participants must be fully ambulatory without the use of a cane, walker, or wheelchair
* Study participants must be able to tolerate moderate aerobic exercise. It will also be required that a physician clear any subjects entering the exercise program who have signs and symptoms suggestive of cardiovascular, cerebrovascular, metabolic, or renal disease and have been active 3 days per week for 30 minutes each day
* Any history of bladder cancer, uterine cancer, ovarian cancer, vaginal cancer, the current placement of a catheter, urethral diverticulum, spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida, cyclophosphamide treatment, radiation cystitis, bladder tuberculosis, or are experiencing an active genital herpes episode
* Pregnant women are not eligible for this study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Interstitial Cystitis Symptom Index (ICSI) Scores | baseline
  Participants answer a series of questions to get a final score. Scores range from 0-20, with 0 being no symptoms and 20 the most severe.
Interstitial Cystitis Problem (ICPI) Index Scores | week 3
  Participants answer a series of questions to get a final score. Scores range from 0-16, with 0 being no symptoms and 16 the most severe.
Interstitial Cystitis Symptom Index (ICSI) Scores | week 3
  Participants answer a series of questions to get a final score. Scores range from 0-20, with 0 being no symptoms and 20 the most severe.
Interstitial Cystitis Problem (ICPI) Index Scores | week 6
  Participants answer a series of questions to get a final score. Scores range from 0-16, with 0 being no symptoms and 16 the most severe.
Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) Scores | baseline
  This survey is used to grade people with chronic pelvic pain. Participants answer a series of questions. Scores range between 0 and 35, and studies have indicated that a score greater than 12 is indicative of significant symptoms
Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) Scores | week 3
  This survey is used to grade people with chronic pelvic pain. Participants answer a series of questions. Scores range between 0 and 35, and studies have indicated that a score greater than 12 is indicative of significant symptoms
Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) Scores | week 6
  This survey is used to grade people with chronic pelvic pain. Participants answer a series of questions. Scores range between 0 and 35, and studies have indicated that a score greater than 12 is indicative of significant symptoms

SECONDARY OUTCOMES:
Change in the Short Form 36 (SF-36) Health Survey Scores | baseline, week 3, week 6
  The SF-36 is a questionnaire that consists of 8 subsections of 36 total questions. The sections are Physical functioning (10 items), Role limitations due to physical health (4 items), Role limitations due to emotional problems (4 items), Energy/fatigue (4 items), Emotional well-being (5 items), Social functioning (2 items), Pain (2 items), General health (5 items). Aggregate scores for each domain range from 0 to 100, compiled as a percentage - where the higher the score, the more favorable the health state of the patient.
Changes in Composite Autonomic Symptom Score (COMPASS-31) Scores | baseline, week 3, week 6
  The test has 6 domains looking at autonomic symptoms: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor. The six domain scores sum to a total COMPASS 31 score of 0 to 100, and a higher COMPASS 31 score indicates more severe autonomic symptoms.

OTHER OUTCOMES:
Changes in inflammatory urinary biomarkers | baseline, 6 weeks
  Urine samples will be obtained at baseline and at the end of the 4 month exercise period from participants. The urine will then be analyzed for biomarkers of inflammation using a Luminex High Performance Assay. Any decrease in the levels of biomarkers of inflammation in the urine is the outcome of interest.
Post-regimen review | after week 6
  After the exercise program concludes, participants will be contacted via phone or email and asked to comment on the program and make suggestions for improvement. This will include things such as if they would recommend the program to friends/family, if they have continued to exercise and/or will continue to exercise on their own time, and any portions of the program they would change or do differently.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Walker, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No